CLINICAL TRIAL: NCT02704299
Title: A Single-centered Clinical Trial of Surgery，Chemotherapy in Combination With Autologous T Cells-Based Immunotherapy for Advanced Gastric Cancer.
Brief Title: The Study of Surgery,Chemotherapy and Autologous T Cells-Based Immunotherapy for Advanced Gastric Cancer.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai AbelZeta Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBMG-TCM-GC-1.1
Record Dates: First submitted 2016-02-26; First posted 2016-03-10 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Gastric Cancer.
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous T cells-Based Immunotherapy (Experimental): Surgery Chemotherapy Autologous T cells-Based Immunotherapy
  Interventions: Biological: Autologous T cells-Based Immunotherapy

INTERVENTIONS:
Biological: Autologous T cells-Based Immunotherapy — TCM cells are the subpopulation of T lymphocytes with key characteristics including high potency and long-term memory of specific immunity.
  Other Names: TCM

SUMMARY:
Evaluate the feasibility ,safety and efficacy of Surgery，Chemotherapy in Combination with Autologous T cells-Based Immunotherapy for Advanced Gastric Cancer.

DETAILED DESCRIPTION:
Safety:AE/SAE Efficacy:immunologic function;FPS

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 80 years, males and females.
* Subjects who understand and sign the consent form for this study.
* The pathologically confirmed advanced gastric cancer T3、T4 or T2 and Metastasis in lymph nodes.
* Subjects are surgical candidates.
* No distant metastasis (M0) and No distant lymph node metastasis.
* Expected survival time of at least 6 months.

Exclusion Criteria:

* Subjects who do not sign the consent form for this study.
* The subject has an allergic history of medicine or food.
* The subject has uncontrolled or hard-to-control diseases of cardiovascular,liver,kidney or lung,endocrine system.
* The subject tests positive for: HIV, hepatitis virus, syphilis or other infectious diseases.
* The subject has an history of other malignant tumour.
* The subject has history of alcoholism, drug abuse, or mental illness in the 12 years prior to this trial.
* The subject has participated in any other clinical trial in the 3 months prior to this trial.
* The subject is pregnant, lactating or planning to conceive within the next 24 months.
* The subject has any other unsuitable or adverse condition to be determined by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival(PFS) | 24months
  The primary objective is to assess progression free survival (PFS).

SECONDARY OUTCOMES:
Incidences of adverse events or serious adverse events | 24months

IPD SHARING:
Plan to Share IPD: Undecided